CLINICAL TRIAL: NCT00215670
Title: A Randomized, Double-Masked, Multi-Center Trial of the Safety, Tolerability and Pharmacokinetics of 1 Mg/Eye and 3 Mg/Eye Intravitreal Injections of Pegaptanib Sodium (Anti-Vegf Pegylated Aptamer) Given Every 6 Weeks for 54 Weeks, in Patients With Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Study of the Safety, Tolerability and Pharmacokinetics of 1 Mg/Eye and 3 Mg/Eye Pegaptanib Sodium in Patients With Exudative Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOP1006
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-05

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Macugen; Pharmacokinetics; Age-Related Macular Degeneration; PK
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

INTERVENTIONS:
Drug: pegaptanib sodium (Macugen)

SUMMARY:
The objectives of this study are to characterize the safety, tolerability and pharmacokinetics of pegaptanib when given as 1 or 3mg/eye intravitreous injections every 6 weeks for 54 weeks in patients with subfoveal choroidal neovascularization (CNV) secondary to AMD.

ELIGIBILITY:
Inclusion Criteria:

Best corrected visual acuity in the study eye between 20/40 and 20/320 and better or equal to 20/800 in the fellow eye.

Subfoveal CNV, secondary to AMD, w/ a total lesion size [including blood, scar/atrophy & neovascularization] of less than or equal to 12 disc areas, of which at least 50% must be active CNV.

Patients of either sex, aged greater than or equal to 50 years.

Exclusion Criteria:

Previous subfoveal thermal laser therapy. Any subfoveal scarring or atrophy & no more than 25% of the total lesion size may be made up of scarring or atrophy.

More than one prior PDT w/ Visudyne is not permitted. Pts may not have rec'd their 1st PDT w/in less than 8 wks or more than 13 wks prior to the BSL angiography/photography for the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2002-11; Study Completion 2006-05